CLINICAL TRIAL: NCT00388193
Title: Burkimab:Study Multicenter of Optimization of the Treatment of LLA-B and the Burkitt's Lymphoma in Adult Patients (From 15 Years Old)
Brief Title: Rituximab Combined With Chemotherapy in Burkitt's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-001067-64
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2013-02

CONDITIONS: Acute Lymphoblastic Leukemia; Burkitt's Lymphoma
Keywords: ALL (L3); BURKITT's LYMPHOMA; RITUXIMAB
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RITUXIMAB

INTERVENTIONS:
Drug: RITUXIMAB — 375 mg/m2/d day 1

SUMMARY:
The purpose of this clinical trial is to prove the efficacy of the following new regimen treatment:

* Administration of anti-CD20 (Rituximab) combined with chemotherapy.
* Combined treatment with high doses of methotrexate and high doses of cytarabine with conventional cytostatics (block C)
* Prophylactic administration of G-CSF after all chemotherapy cycles
* local irradiation after 6 cycle if CNS was affected or if there are residual tumour

DETAILED DESCRIPTION:
Clinical Trial with a pharmaceutical speciality in new conditions to use.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mature LLA-B cell (LLA-L3)
* Patients diagnosed with Burkitt´s and Burkitt´s Like Lymphoma
* Patients 15 years old or up
* Written Informed Consent signed

Exclusion Criteria:

* Serious complications related with LAL3/LB or Secondary illness:

Serious complications, uncontrollable, for example, sepsis, pneumonia with hypoxia, shock, haemorrhage at diagnosis.

* Renal failure unconditional for the Lymphoma/Leukemia
* Heart failure or serious liver.
* Pulmonary obstructive disease or serious restrictive that not allow to treat the patient with intensive chemotherapy.
* Secondary Lymphoma after chemotherapy or previous radiotherapy or second malignant tumour.
* Known hypersensitivity to any foreign protein.
* Previous treatment with cytostatics of the LLA-B or Burkitt´s Lymphoma (exception: administration on short time of glucocorticoids ≤ 7 days, one administration of vincristine or cyclophosphamide, one cycle of CHOP, urgent administration of the another cytostatics).
* With another malignant tumour in the last 5 year.
* Women in fertile age must give positive in the pregnancy test or nursing mother.
* Mental disability or emotional or psychiatric significant disorder were the patient can't understand nor cooperate with treatment.
* Patients is enrolled in another clinical research study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Determinate the efficacy of the administration of anti-CD20 (RITUXIMAB) combined with chemotherapy. | 1 year

SECONDARY OUTCOMES:
Combined treatment with high doses of methotrexate and high doses of cytarabine with conventional cytostatics (block C) | 1 year
Prophylactic administration of G-CSF after all chemotherapy cycles | 1 year
local irradiation after 6 cycle if CNS was affected or if there are residual tumour | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ribera Josep Mª, Dr, Study Chair — Germans Trias i Pujol Hospital
Locations (15):
- Spain (15):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital "Santa Creu i Sant Pau", Barcelona, Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Universitario Morales Meseguer, Murcia, Murcia, Murcia
  - Hospital Carlos Haya, Málaga, Málaga
  - Hospital Son Dureta, Palma de Mallorca, Palma de Mallorca
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital La Fe, Valencia, Valencia
  - Complejo Hospitalario de Cáceres, Cáceres
  - Hospital general de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Txagorritxu, Vitoria-Gasteiz

REFERENCES:
- [Background] Hoelzer D, Ludwig WD, Thiel E, Gassmann W, Loffler H, Fonatsch C, Rieder H, Heil G, Heinze B, Arnold R, Hossfeld D, Buchner T, Koch P, Freund M, Hiddemann W, Maschmeyer G, Heyll A, Aul C, Faak T, Kuse R, Ittel TH, Gramatzki M, Diedrich H, Kolbe K, Fuhr HG, Fischer K, Schadeck-Gressel C, Weiss A, Strohscheer I, Metzner B, Fabry U, Gokbuget N, Volkers B, Messerer D, Uberla K. Improved outcome in adult B-cell acute lymphoblastic leukemia. Blood. 1996 Jan 15;87(2):495-508. PMID 8555471
- [Background] Reiter A, Schrappe M, Tiemann M, Ludwig WD, Yakisan E, Zimmermann M, Mann G, Chott A, Ebell W, Klingebiel T, Graf N, Kremens B, Muller-Weihrich S, Pluss HJ, Zintl F, Henze G, Riehm H. Improved treatment results in childhood B-cell neoplasms with tailored intensification of therapy: A report of the Berlin-Frankfurt-Munster Group Trial NHL-BFM 90. Blood. 1999 Nov 15;94(10):3294-306. PMID 10552938
- [Background] Thomas DA, Cortes J, O'Brien S, Pierce S, Faderl S, Albitar M, Hagemeister FB, Cabanillas FF, Murphy S, Keating MJ, Kantarjian H. Hyper-CVAD program in Burkitt's-type adult acute lymphoblastic leukemia. J Clin Oncol. 1999 Aug;17(8):2461-70. doi: 10.1200/JCO.1999.17.8.2461. PMID 10561310
- [Background] Adde M, Shad A, Venzon D, Arndt C, Gootenberg J, Neely J, Nieder M, Owen W, Seibel N, Wilson W, Horak ID, Magrath I. Additional chemotherapy agents improve treatment outcome for children and adults with advanced B-cell lymphomas. Semin Oncol. 1998 Apr;25(2 Suppl 4):33-9; discussion 45-8. PMID 9578060
- [Background] Mounier N, Briere J, Gisselbrecht C, Emile JF, Lederlin P, Sebban C, Berger F, Bosly A, Morel P, Tilly H, Bouabdallah R, Reyes F, Gaulard P, Coiffier B. Rituximab plus CHOP (R-CHOP) overcomes bcl-2--associated resistance to chemotherapy in elderly patients with diffuse large B-cell lymphoma (DLBCL). Blood. 2003 Jun 1;101(11):4279-84. doi: 10.1182/blood-2002-11-3442. Epub 2003 Feb 6. PMID 12576316
- [Background] Lee EJ, Petroni GR, Schiffer CA, Freter CE, Johnson JL, Barcos M, Frizzera G, Bloomfield CD, Peterson BA. Brief-duration high-intensity chemotherapy for patients with small noncleaved-cell lymphoma or FAB L3 acute lymphocytic leukemia: results of cancer and leukemia group B study 9251. J Clin Oncol. 2001 Oct 15;19(20):4014-22. doi: 10.1200/JCO.2001.19.20.4014. PMID 11600602
- [Background] Zinzani PL, Martelli M, Magagnoli M, Pescarmona E, Scaramucci L, Palombi F, Bendandi M, Martelli MP, Ascani S, Orcioni GF, Pileri SA, Mandelli F, Tura S. Treatment and clinical management of primary mediastinal large B-cell lymphoma with sclerosis: MACOP-B regimen and mediastinal radiotherapy monitored by (67)Gallium scan in 50 patients. Blood. 1999 Nov 15;94(10):3289-93. PMID 10552937
- [Background] Oriol A, Ribera JM, Esteve J, Sanz MA, Brunet S, Garcia-Boyero R, Fernandez-Abellan P, Marti JM, Abella E, Sanchez-Delgado M, Penarrubia MJ, Besalduch J, Moreno MJ, Borrego D, Feliu E, Ortega JJ; PETHEMA Group, Spanish Society of Hematology. Lack of influence of human immunodeficiency virus infection status in the response to therapy and survival of adult patients with mature B-cell lymphoma or leukemia. Results of the PETHEMA-LAL3/97 study. Haematologica. 2003 Apr;88(4):445-53. PMID 12681972
- See also: Spanish association of Haematology — http://www.aehh.org